CLINICAL TRIAL: NCT01579656
Title: The Effects of Four Commonly Consumed Seeds (Flax, Poppy, Sesame & Salba) on Postprandial Blood Glucose Response, Vascular, Appetite and Sensory Parameters in Healthy Individuals
Brief Title: Effect of Flax, Poppy, Sesame & Salba on Postprandial Blood Glucose Response, Vascular, Appetite & Sensory Parameters
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Vladimir Vuksan, Dr. Vladimir Vuksan, Unity Health Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: GLUSEED-2
Record Dates: First submitted 2011-08-26; First posted 2012-04-18 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — S-adenosyl-L-methionine (R,S)-reticuline 7-O-methyltransferase; Linseed Oil; Dietary Fiber

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Salba (Experimental): 25g of ground Salba baked into a bran muffin
  Interventions: Dietary Supplement: Salba
- Poppy (Experimental): 25g of ground poppy seeds baked into a bran muffin
  Interventions: Dietary Supplement: Poppy
- Flaxseed (Experimental): 25g of ground flaxseed baked into a bran muffin
  Interventions: Dietary Supplement: Flaxseed
- Sesame (Experimental): 25g of ground sesame seeds baked into a bran muffin
  Interventions: Dietary Supplement: Sesame
- Wheat Bran (Placebo Comparator): Bran muffin matched for total available carbohydrates, total dietary fibre and calories
  Interventions: Dietary Supplement: Wheat Bran

INTERVENTIONS:
Dietary Supplement: Salba — 25g of ground Salba baked into a bran muffin matched for total available carbohydrate (50g), total dietary fibre (15g), and calories (494.5 kcal) with the addition of flour, inulin or canola oil. One of five muffins (Salba, Poppy, Sesame, Flax, Bran) will be administered at each visit.
  Other Names: Salba hispanica L.
  Arms: Salba
Dietary Supplement: Poppy — 25g of ground Poppy Seeds baked into a bran muffin matched for total available carbohydrate (50g), total dietary fibre (15g), and calories (494.5 kcal) with the addition of flour, inulin or canola oil. One of five muffins (Salba, Poppy, Sesame, Flax, Bran) will be administered at each visit.
  Other Names: Papaver somniferum L.
  Arms: Poppy
Dietary Supplement: Flaxseed — 25g of ground Flaxseed baked into a bran muffin matched for total available carbohydrate (50g), total dietary fibre (15g), and calories (494.5 kcal) with the addition of flour, inulin or canola oil. One of five muffins (Salba, Poppy, Sesame, Flax, Bran) will be administered at each visit.
  Other Names: Linum Usitatissimum
  Arms: Flaxseed
Dietary Supplement: Sesame — 25g of ground Sesame Seeds baked into a bran muffin matched for total available carbohydrate (50g), total dietary fibre (15g), and calories (494.5 kcal) with the addition of flour, inulin or canola oil. One of five muffins (Salba, Poppy, Sesame, Flax, Bran) will be administered at each visit.
  Other Names: Sesamum indicum
  Arms: Sesame
Dietary Supplement: Wheat Bran — Bran muffin matched for total available carbohydrate (50g), total dietary fibre (15g), and calories (494.5 kcal). One of five muffins (Salba, Poppy, Sesame, Flax, Bran) will be administered at each visit.
  Other Names: Quaker Bran Muffin Mix
  Arms: Wheat Bran

SUMMARY:
Consumption of whole grains has been heavily endorsed by both government and major health agencies, as evidenced in Health Canada's Food Guide, the US Department of Agriculture's Food Pyramid, and the Heart and Stroke Foundation's healthy eating guide. Whole grains have been championed for their proposed cardioprotective and weight control effects as suggested by epidemiological studies. The health benefits of whole grain products may be attributable to their nutrient composition, which contains dietary fibre, protein and several essential nutrients. There has also been a concurrent increase in seed consumption. Seeds have a similar and potentially superior nutritional composition to whole grains and they are rich in mammalian lignans and polyunsaturated fats, especially the highly valued omega-3 fatty acids. Preliminary studies on seeds have shown that they impart health benefits similar to those imparted by whole grains. Consumer choices regarding seed consumption may be based on their potential health benefits. Furthermore, they may also be affected by subjective sensory factors, such as appearance, taste and pre-conceived perceptions. Therefore, this study will compare the health properties of four seeds and their effects on appetite and sensory parameters in healthy individuals. These four seeds will be that of flax, poppy and sesame, due to their popularity and consumption as well as Salba, which has also recently received much attention for its associated health benefits.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years
* normal glycemic response
* BMI between 18.5 - 25 kg/m2
* peripheral systolic and diastolic blood pressure < 140mmHg and < 90mmHg

Exclusion Criteria:

* known history of liver or kidney disease, diabetes, hypertension, stroke or myocardial infarctions, thyroid disease, Celiac disease/gastrointestinal disease, or AIDS;
* allergies to any of the test products
* using prescription medications or Natural Health Products
* any condition which, in the opinion of the investigator, might jeopardize the health and safety of the subject or study personnel, or adversely affect the study results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-02; Primary Completion 2012-04 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Postprandial Blood Glucose | 3 hours
  At each visit, postprandial blood glucose will be measured every 15 minutes over 3 hours.

SECONDARY OUTCOMES:
Blood Pressure | 3 hours
  At each visit, brachial blood pressure will be measured every 30 minutes over 3 hours.
Arterial Stiffness | 3 hours
  At each visit, arterial stiffness (assessed by central augmentation index) will be measured every 30 minutes over 3 hours.
Palatability | 3 hours
  At each visit, participants will record their subjective ratings using a 100mm visual analogue scale and these ratings will be combined into a total subjective palatability score.
Personal Preference | 3 hours
  At each visit, participants will record their subjective ratings using a 100mm visual analogue scale and these ratings will be combined into a total subjective personal preference score.
Satiety | 3 hours
  At each visit, participants will record their subjective ratings using a 100mm visual analogue scale and these ratings will be combined into a total subjective appetite score.

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Vuksan, PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada